CLINICAL TRIAL: NCT00130442
Title: A Phase II Study of PI-88 With Dacarbazine in Patients With Metastatic Melanoma
Brief Title: Trial of PI-88 With Dacarbazine in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cellxpert Biotechnology Corp. (Industry)
Collaborators: Medigen Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR88205; NCT00128648 (obsolete NCT alias)
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Melanoma
Keywords: phase II; metastatic melanoma; dacarbazine; combination; PI-88
MeSH Terms: conditions — Melanoma | interventions — phosphomannopentaose sulfate; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1- PI-88 plus dacarbazine (Experimental): PI-88 (muparfostat) 190 mg daily by subcutaneous injection and dacarbazine 1000 mg/m2 on day 1 of each 21 day cycle
  Interventions: Drug: PI-88 and dacarbazine
- Arm 2- dacarbazine alone (Active Comparator): dacarbazine 1000 mg/m2 on day 1 of every 21 day cycle by intravenous infusion
  Interventions: Drug: dacarbazine or DTIC

INTERVENTIONS:
Drug: PI-88 and dacarbazine — 190 mg daily by subcutaneous injection for PI-88 and 1000 mg/m2 on day 1 of each 21 day cycle by intravenous infusion
  Arms: Arm 1- PI-88 plus dacarbazine
Drug: dacarbazine or DTIC — intravenous infusion 1000 mg/m2 on day 1 of every 21 day cycle
  Arms: Arm 2- dacarbazine alone

SUMMARY:
The aim of the study is to compare the safety and effectiveness of a new drug called PI-88, when used in combination with an approved chemotherapy drug called dacarbazine, in the treatment of metastatic melanoma.

PI-88 blocks new blood vessel growth in tumours (starves it of nutrients) and dacarbazine stops the cancer cells from growing. The results from this study will be analysed to see if it is worthwhile for the two drugs to be tested in future studies involving larger numbers of melanoma patients.

DETAILED DESCRIPTION:
Metastatic melanoma is a difficult-to-treat cancer for which available treatment options are limited and minimally effective. Dacarbazine is currently one of the standard chemotherapy drugs used for the treatment of metastatic melanoma. However, it is associated with low response rates (10-20%) and median survival of less than 12 months (6-11 months in most studies). PI-88 is an antiangiogenic and antimetastatic drug that has already shown some evidence of efficacy when used alone in an intermittent dosage regimen (4 consecutive days per week) in the treatment of patients with advanced melanoma. The FDA has designated PI-88 as an Orphan Drug for this indication, as well as for Stage III and high-risk stage II disease. The aim of this randomised pilot phase II trial is to determine whether PI-88 in combination with a standard regimen of dacarbazine (1000 mg/m2 every 3 weeks) should be considered for further investigation in a larger-scale trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven metastatic melanoma
* Surgery not feasible or inappropriate
* Measurable disease. Metastatic lesions must be measurable by magnetic resonance imaging (MRI) or computed tomography (CT) as defined in Response Evaluation Criteria in Solid Tumors (RECIST), and cutaneous lesions by physical examination.
* Have voluntarily given written informed consent to participate in this study
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1
* Life expectancy at least 3 months
* Neutrophil count > 1.5 x 10^9/L (1,500/mm3)
* Platelet count > 100 x 10^9/L (100,000/mm3)
* Acceptable liver function tests (see Exclusion Criteria for maximum allowable elevations of ALT, AST, ALP and LDH)
* PT < 1.5 x upper limit of normal (ULN)
* APTT < 1.5 x ULN
* Creatinine clearance > 40 mL/min, calculated using the Cockcroft-Gault formula (if just below 40 mL/min, then GFR > 40 mL/min as determined by 24-hour urine collection)

Exclusion Criteria:

* Current or history of central nervous system involvement, brain or meningeal metastases
* Ocular melanoma
* Clinically significant non-malignant disease
* Prior or co-existent malignancies (other than stage I internal malignancy where treated and disease-free for > 5 years, non-melanomatous skin cancer or in situ cancer of the cervix)
* Prior chemotherapy
* Prior treatment with vaccines and/or biological response modifiers within the previous 4 weeks
* Prior treatment with radiotherapy within the previous 4 weeks (local palliative radiotherapy is permitted)
* Radiotherapy to > 30% of marrow-bearing bone within the previous 3 months
* Major surgery within the past 4 weeks
* Concomitant use of aspirin (> 150 mg/day), non-steroidal anti-inflammatory drugs (except specific COX-2 inhibitors), heparin, low molecular weight heparin, warfarin (> 1 mg/day) or anti-platelet drugs (abciximab, clopidogrel, dipyridamole, ticlopidine and tirofiban). Low-dose aspirin (≤ 150 mg/day) and low-dose warfarin (≤ 1 mg/day) are permitted as concomitant medications.
* Heparin or low molecular weight heparin within the previous 2 weeks
* History of acute or chronic gastrointestinal bleeding within the last 2 years, inflammatory bowel disease or other abnormal bleeding tendency
* Patients at risk of bleeding due to open wounds or planned surgery
* Bilirubin > 1.5 x ULN
* AST or ALT > 3 x ULN unless patient has hepatic metastases
* LDH > 2 x ULN
* Alkaline phosphatase > 5 x ULN, unless patient has bone metastases
* Myocardial infarction, stroke or congestive heart failure within the past 3 months
* Women who are pregnant or breast feeding
* Women of childbearing potential in whom pregnancy cannot be excluded or who are not using an adequate method of contraception
* History of allergy and/or hypersensitivity to anti-coagulants/thrombolytic agents, especially heparin
* History of immune-mediated thrombocytopenia, thrombotic thrombocytopenic purpura or other platelet disease, or laboratory evidence of anti-heparin antibodies
* Uncontrolled or serious infection within the past 4 weeks
* Patients who are unable to be compliant or to follow instructions given to them by clinic staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2005-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Millward, MD, Study Chair — Sir Charles Gairdner Hospital; Anne Hamilton, PhD, Principal Investigator — Sydney Cancer Centre; Damien Thomson, MD, Principal Investigator — Princess Alexandra Hospital
Locations (12):
- United States (3):
  - Arizona Cancer Centre, Tucson, Arizona
  - University of Colorado Health Science Centre, Denver, Colorado
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
- Australia (9):
  - Sydney Cancer Centre, Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Westmead Institute for Cancer Research, Sydney, New South Wales
  - Wesley Research Institute, Auchenflower, Queensland
  - Townsville Cancer Centre, Townsville, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Border Medical Oncology, Wodonga, Victoria
  - Royal Perth Hospital, Perth, Western Australia
  - Sir Charles Gairdner Hospital, Perth, Western Australia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1- PI-88 Plus Dacarbazine | Arm 2- Dacarbazine Alone
Started | 66 | 68
Completed | 65 | 66
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — did not meet criteria | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population, defined as subjects who received at least one dose of study drug/s
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1- PI-88 Plus Dacarbazine | Arm 2- Dacarbazine Alone | Total
Number analyzed (Participants) | 65 | 66 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (13.26) | 57.9 (13.07) | 59.1 (13.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 27 | 42
  Male | 50 | 39 | 89
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 63 | 65 | 128
  Other | 2 | 1 | 3
Height [Mean (Standard Deviation); unit: cm] | 174.0 (8.11) | 171.2 (9.57) | 172.6 (8.95)
Weight [Mean (Standard Deviation); unit: kg] | 85.11 (15.46) | 81.54 (17.25) | 83.31 (16.42)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.15 (5.277) | 27.64 (5.100) | 27.89 (5.175)
ECOG status [Number; unit: participants] — The ECOG Performance Status is used to assess the functional status in terms of their ability to care for themselves, daily activity, and physical ability. ECOG uses 5 points score from grade 0 to grade 5, where lower grade indicates better independence.
  participants
    0 | 44 | 45 | 89
    1 | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Non-progression Rate After Six Cycles
Description: The Proportion of Patients With Objective Response or Stable Disease (Non-progression Rate) after six treatment cycles
Time Frame: In week 3 of every second cycle (each cycle was 21 days) for all subjects enrolled, up to the end of cycle 6 (About 5 months after randomization)
Population: ITT population consisted of all subjects randomised to treatment who received at least one dose of study medication, had a valid baseline measurement and who had returned for at least one visit post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1- PI-88 Plus Dacarbazine | Arm 2- Dacarbazine Alone
Number analyzed (Participants) | 65 | 65
Participants
  Non-progressed | 13 | 18
  Progressed | 52 | 47

2. Secondary Outcome: Non-progression Rate
Description: The Proportion of Patients With Objective Response or Stable Disease (Non-progression Rate) after 2 or 4 treatment cycles
Time Frame: In week 3 of every second cycle (each cycle was 21 days) for all subjects enrolled in cycle 2 and cycle 4.
Population: ITT population, consisted of all subjects randomised to treatment who received at least one dose of study medication, had a valid baseline measurement and who had returned for at least one visit post-baseline.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1- PI-88 Plus Dacarbazine: PI-88 (muparfostat) 190 mg daily by subcutaneous injection and dacarbazine 1000 mg/m2 on day 1 of each 21 day cycle PI-88 and dacarbazine: 190 mg daily by subcutaneous injection for PI-88 and 1000 mg/m2 on day 1 of each 21 day cycle by intravenous infusion
- Arm 2- Dacarbazine Alone: dacarbazine 1000 mg/m2 on day 1 of every 21 day cycle by intravenous infusion dacarbazine or DTIC: intravenous infusion 1000 mg/m2 on day 1 of every 21 day cycle
Arm/Group | Arm 1- PI-88 Plus Dacarbazine | Arm 2- Dacarbazine Alone
Number analyzed (Participants) | 65 | 65
Participants
  End of cycle 2_Non-progressed | 33 | 35
  End of cycle 2_progressed | 32 | 30
  End of cycle 4_Non-progressed | 24 | 31
  End of cycle 4_progressed | 41 | 33

3. Secondary Outcome: Time to Progression
Description: treatment was to continue until the subject experienced disease progression.
Time Frame: At screening and in week 3 of every second cycle up to the end of cycle 6 and every third cycle after cycle 6 . Each cycle was 21 days.Assessed from date of randomization until the date of first documented progression, up to 50 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm 1- PI-88 Plus Dacarbazine | Arm 2- Dacarbazine Alone
Number analyzed (Participants) | 65 | 65
days | 66 [43 to 134] | 82 [43 to 187]

4. Secondary Outcome: Duration of Response
Description: time from commencement to radiological evidence of progression
Time Frame: At screening and in week 3 of every second cycle up to the end of cycle 6 and every third cycle after cycle 6. Each cycle was 21 days. Assessed from date of randomization until the date of first documented progression, up to 50 months.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1- PI-88 Plus Dacarbazine | Arm 2- Dacarbazine Alone
Number analyzed (Participants) | 65 | 65
days | 117.0 (65.73) | 140.6 (89.38)

5. Secondary Outcome: Survival
Description: time to death and also at time-points 6 month and 12 months
Time Frame: It was to assess time to death. The time frame is at least 6th month, 12th month and data was continuously collected till the end of the study, up to 50 months..
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm 1- PI-88 Plus Dacarbazine | Arm 2- Dacarbazine Alone
Number analyzed (Participants) | 65 | 65
days | 304.00 [224.00 to 366.00] | 416.00 [304.00 to 476.00]

ADVERSE EVENTS:
Arm/Group | Arm 1- PI-88 Plus Dacarbazine | Arm 2- Dacarbazine Alone
Serious Adverse Events (participants affected / at risk) | 20/65 | 13/66
Other Adverse Events (participants affected / at risk) | 65/65 | 61/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1- PI-88 Plus Dacarbazine (N=65) | Arm 2- Dacarbazine Alone (N=66)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Antibody test positive (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1- PI-88 Plus Dacarbazine (N=65) | Arm 2- Dacarbazine Alone (N=66)
Neutropenia (Blood and lymphatic system disorders) | 20 | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 15 | 8
Palpitations (Cardiac disorders) | 4 | 1
Visual impairment (Eye disorders) | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 9
Constipation (Gastrointestinal disorders) | 25 | 16
Diarrhoea (Gastrointestinal disorders) | 14 | 16
Dry mouth (Gastrointestinal disorders) | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 7 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 4
Nausea (Gastrointestinal disorders) | 35 | 39
Vomiting (Gastrointestinal disorders) | 14 | 13
Chest pain (General disorders) | 7 | 8
Chills (General disorders) | 3 | 7
Fatigue (General disorders) | 39 | 39
Infusion site pain (General disorders) | 4 | 8
Injection site haematoma (General disorders) | 30 | 1
Inject site pain (General disorders) | 14 | 2
Injection site reaction (General disorders) | 12 | 0
Oedema peripheral (General disorders) | 6 | 2
Pain (General disorders) | 4 | 5
Pyrexia (General disorders) | 3 | 8
Lower respiratory track infection (Infections and infestations) | 2 | 5
Nasopharyngitis (Infections and infestations) | 3 | 7
Upper respiratory tract infection (Infections and infestations) | 4 | 6
Contusion (Injury, poisoning and procedural complications) | 13 | 5
Alanine aminotransferase increased (Investigations) | 6 | 0
Platelet count decreased (Investigations) | 4 | 0
Weight decreased (Investigations) | 4 | 3
Decreased appetite (Metabolism and nutrition disorders) | 14 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 1
Burning sensation (Nervous system disorders) | 5 | 0
Dizziness (Nervous system disorders) | 14 | 13
Dysgeusia (Nervous system disorders) | 4 | 4
Headache (Nervous system disorders) | 11 | 16
Lethargy (Nervous system disorders) | 7 | 3
Anxiety (Psychiatric disorders) | 4 | 2
Depression (Psychiatric disorders) | 2 | 7
Insomnia (Psychiatric disorders) | 16 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 4
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 3 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 3
Rash (Skin and subcutaneous tissue disorders) | 7 | 6
Flushing (Vascular disorders) | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No